CLINICAL TRIAL: NCT06850896
Title: Effects of Early Antibiotic Exposure on Gut Microbiota and Motility Establishment in Newborns: a Prospective Cohort Study
Brief Title: Antibiotic Exposure on Gut Microbiota and Motility Establishment in Newborns
Status: Active, not recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: 25K041-001
Record Dates: First submitted 2025-02-26; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: NEC - Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Preterm Infants with Antibiotic Exposure: Description: Newborns with gestational age 24-36 weeks who receive antibiotics within the first 72 hours of life.

SUMMARY:
This prospective cohort study aims to investigate the impact of early antibiotic exposure on the establishment of gut microbiota and motility in newborns, particularly preterm infants. The study will explore the correlation between antibiotic exposure, gut microbiota colonization, and 5-hydroxytryptamine (5-HT) levels, which are critical for gastrointestinal motility. The findings may provide insights into optimizing antibiotic use and improving gastrointestinal health in neonates.

ELIGIBILITY:
Inclusion Criteria:

* Newborns admitted within 72 hours of birth
* Gestational age 24-36 weeks (preterm) and term infants
* Informed consent obtained from parents or guardian

Exclusion Criteria:

* Congenital gastrointestinal malformations (e.g., intestinal atresia, Hirschsprung's disease)
* Severe systemic or organ-specific diseases
* Expected mortality due to severe illness

Ages: 24 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will enroll newborns admitted to the neonatal unit of Jilin University First Hospital from November 2024 to November 2027.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
gut microbiota | Enrollment Period: This is the time during which participants will be recruited and enrolled into the study. You have specified that enrollment will occur from November 2024 to November 2027. Intervention Period: Since this is an observational study, the
  Impact of antibiotic exposure on gut microbiota colonization assessed by 16S rRNA sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin university, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang S, Zhang L, Yan W, Li S, Han J, Zhou Q, Yang Y, Lee SK, Cao Y; REIN-EPIQ Study Group. Antibiotic Use in Neonatal Intensive Care Units in China: A Multicenter Cohort Study. J Pediatr. 2021 Dec;239:136-142.e4. doi: 10.1016/j.jpeds.2021.08.067. Epub 2021 Aug 28. PMID 34461063